CLINICAL TRIAL: NCT03893994
Title: Effect Of Stretching Programme On Shoulder Performance In Volleyball Players With Posterior Shoulder Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Irem Duzgun, Principal Investigator, PT, PhD, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 1817KA-17141
Record Dates: First submitted 2019-03-14; First posted 2019-03-28 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Posterior Shoulder Tightness
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stretching group (Experimental): Posterior shoulder stretching exercises
  Interventions: Other: Stretching exercises
- Control Group (No Intervention): No exercise will be applied

INTERVENTIONS:
Other: Stretching exercises — Stretching exercises will be applied 6 days a week, 30sec / 5 reps
  Arms: Stretching group

SUMMARY:
When the dominant arm is compared with the non-dominant arm in overhead athletes there is a serious internal rotation limitation in the dominant arm. Due to overhead activity, adaptive changes in shoulder joint mobility and flexibility are indicated. Internal rotation limitation is often associated with increased external rotation. One of the reason of this adaptive change is posterior shoulder tightness which is common in overhead athletes as well as in volleyball players. The aim of this study is to determine the effect of stretching program on the range of motion, flexibility of posterior shoulder muscles and functional performance.

ELIGIBILITY:
Inclusion Criteria:

* Posterior shoulder tightness ( 15 degree internal rotation limitation compared with non dominant side)
* Being a professional volleyball player ( at least 3 years experience in the professional league)
* At least having 4 training days in a week
* negative impingement tests ( Hawkins, Neer or Jobe)
* No shoulder pain

Exclusion Criteria:

* Having any shoulder surgery
* Having a shoulder injury in last 6 months
* Having any neck problem or neck pain
* Having a systemic illness
* Sublocated shoulder

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in shoulder internal ROM measurement with digital inclometery at 6 weeks | 6 weeks
  Passive shoulder internal rotation gain which is measured with digital inclometery

SECONDARY OUTCOMES:
Mean change from baseline in muscle hardness (kPA) with elastography at 6 weeks | 6 weeks
  Elastrography will be used to measure muscle hardness (kPA)
Mean change from baseline in distance scores on single arm shot put test at 6 weeks | 6 weeks
  Single arm shot put test will be used to assess arm power. Distance will be measured in cm.
Mean change from baseline in velocity (km/h) of spike with radar at 6 weeks | 6 weeks
  Spike velocity will be measured with radar (km/h)
Mean change from baseline in strength ( Nm/kg) of shoulder internal rotation and external rotation at 6 weeks | 6 weeks
  Isokinetic measurements of internal and external shoulder rotation (Nm/kg) at 60 degree/ Sec and 180 degree/ Sec speed will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- Turkish Volleyball Federation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No